CLINICAL TRIAL: NCT02814188
Title: Effects of Pre-Exercise Nutrition Strategies on Body Temperature and Thermoregulatory Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Patrick Wilson, PhD, Assistant Professor of Exercise Science, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 892213-3
Record Dates: First submitted 2016-06-20; First posted 2016-06-27 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Impaired Thermoregulation
Keywords: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbohydrate Beverage (Experimental)
  Interventions: Other: Carbohydrate Beverage
- Placebo Beverage (Placebo Comparator)
  Interventions: Other: Placebo Beverage

INTERVENTIONS:
Other: Carbohydrate Beverage — 750 ml of a 13.5% carbohydrate (sucrose) beverage
  Arms: Carbohydrate Beverage
Other: Placebo Beverage — 750 ml of an artificially-sweetened beverage
  Arms: Placebo Beverage

SUMMARY:
Carbohydrate ingestion, in particular fructose, has been shown in a handful of previous studies to elicit a thermic effect and increase core body temperature after ingestion. Carbohydrate foods and supplements are commonly consumed prior to endurance running competition, including situations where an athlete's ability to dissipate body heat is compromised. Thus, there is some potential for pre-exercise carbohydrate ingestion to have a deleterious effect on body heat regulation in hot and humid environments. Thus, this projects aims to study the effects of pre-exercise carbohydrate ingestion on core body temperature, perceived thermal stress, and perceived exertion during high-intensity running.

ELIGIBILITY:
Inclusion Criteria:

* Be currently running ≥20 miles per week
* Have a projected 5-km maximal effort running time between 16:00-23:00 minutes

Exclusion Criteria:

* Any gastrointestinal disorders that cause swallowing problems or frequent nausea/vomiting

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-06; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Core Body Temperature | 80 minutes (60, 50, 40, 30, 20, and 10 min pre-run and at 1-km intervals during a 20 min 5-km run)
  Core body temperature will be measured with a ingestible pill thermometer. Readings will be taken during a 60 minute rest period and at 1-km intervals during a 5-km run.

SECONDARY OUTCOMES:
Thermal Sensation Scale | 80 minutes (60, 50, 40, 30, 20, and 10 min pre-run and at 1-km intervals during a 20 min 5-km run)
  The Thermal Sensation Scale is a 0-8 numerical rating scale with descriptors of "unbearably cold" at 0, "neutral" at 4, and "unbearably hot" at 8. These ratings will be collected during a 60 minute rest period and at 1-km intervals during a 5-km run.
Feeling Scale | 80 minutes (60, 50, 40, 30, 20, and 10 min pre-run and at 1-km intervals during a 20 min 5-km run)
  The Feeling Scale is a bipolar numerical rating scale ranging from -5 to +5, with descriptors of "very bad" at -5, "neutral" at 0, and "very good" at +5. These ratings will be collected during a 60 minute rest period and at 1-km intervals during a 5-km run.
Rating of Perceived Exertion | 80 minutes (60, 50, 40, 30, 20, and 10 min pre-run and at 1-km intervals during a 20 min 5-km run)
  These ratings will be collected during a 60 minute rest period and at 1-km intervals during a 5-km run.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Performance Laboratory, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No